CLINICAL TRIAL: NCT04590287
Title: The Use of ICF Classification System in Secondary Prevention of Cardiovascular Disease Among Others Ischemic and Hemorrhagic Stroke.
Brief Title: ICF in Secondary Prevention of Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 4/2020
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Cardiovascular Diseases; Secondary Prevention; Risk Factor, Cardiovascular
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients after ischemic stroke: The analysis included the presence of CVD risk factors in patients after ischemic stroke durning in the early rehabilitation.
- Patients after hemorrhagic stroke: The analysis included the presence of CVD risk factors in patients after hemorrhagic stroke durning in the early rehabilitation.

SUMMARY:
The aim of this study was to develop a practical protocol based on the ICF(The International Classification of Functioning, Disability, and Health) the risk factors of cardiovascular disease (CVD) in secondary prevention.

DETAILED DESCRIPTION:
The original ICF assessment sheet contains CVD risk factor categories, such as comorbidities (depressive disorders, insomnia, heart rhythm and heart rate disorders, carotid artery disease, and hypertension), measures of liver and renal impairment, disorders of carbohydrate and lipid metabolism). The evaluation criteria for each category were determined based on recommendations defined in the ESC, AHA, EFSD, and KIDIGO guidelines.

ELIGIBILITY:
Inclusion Criteria:

* the first episode of ischemic stroke or hemorrhagic stroke,
* full medical documentation with a description of the above-mentioned risk factors

Exclusion Criteria:

* another neurological disease: brain tumor, trauma craniocerebral
* incomplete medical history - no data on assessed risk factors CVD

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients after ischemic stroke 60 patients after hemorrhagic stroke
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
emotional functions | first examination on admission
  symptoms of depression
sleep functions | first examination on admission
  symptoms of insomnia
heart rate | first examination on admission
  heart rate per minute
heart rhythm | first examination on admission
  heart rhythm interpreting ECG (regular or irregular)
functions of arteries | first examination on admission
  carotid stenosis [%]
increased blood pressure | first examination on admission
  blood pressure value [mm/Hg]
functions related to the coagulation of blood. | first examination on admission
  International Normalised Ratio (INR) testing
Glycosylated hemoglobin | first examination on admission
  HbA1c [%]
lipid metabolism. | first examination on admission
  LDL [mg/dL]

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Chlebuś, MD, Principal Investigator — Clinic Rehabilitation, University of Medical Sciences in Poznań
Locations (1):
- Department of Rehabilitation and Physiotherapy Rehabilitation,, Poznan, Poland

REFERENCES:
- [Derived] Lucki M, Chlebus E, Warenczak A, Lisinski P. Risk Factors for the Recurrence of CVD Incidents in Post-Stroke Patients over a 5-Year Follow-Up Period Based on the ICF Classification. Int J Environ Res Public Health. 2021 Jun 3;18(11):6021. doi: 10.3390/ijerph18116021. PMID 34205106